CLINICAL TRIAL: NCT02547922
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Phase 2 Study Evaluating the Efficacy and Safety of Anifrolumab in Adult Subjects With Active Proliferative Lupus Nephritis
Brief Title: Safety and Efficacy of Two Doses of Anifrolumab Compared to Placebo in Adult Subjects With Active Proliferative Lupus Nephritis
Acronym: TULIP-LN1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3461C00007
Record Dates: First submitted 2015-08-31; First posted 2015-09-14 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Lupus Nephritis
Keywords: lupus, nephritis, randomized, placebo, anifrolumab, safety, efficacy, adult
MeSH Terms: conditions — Lupus Nephritis; Nephritis | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Anifrolumab - Lower Dose (Experimental): Anifrolumab - Lower Dose
  Interventions: Biological: Anifrolumab
- Anifrolumab - Higher Dose (Experimental): Anifrolumab - Higher Dose
  Interventions: Biological: Anifrolumab
- Placebo (Placebo Comparator): Placebo IV Q4W plus SOC
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Anifrolumab — Administration every 4 week from Week 0 to Week 100 in addition to SOC which will continue until Week 112
  Arms: Anifrolumab - Higher Dose; Anifrolumab - Lower Dose
Drug: Placebo — Administration every 4 week from Week 0 to Week 100 in addition to SOC which will continue until Week 112
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an intravenous treatment regimen of two doses of anifrolumab versus placebo in adult subjects with active proliferative lupus nephritis (LN).

DETAILED DESCRIPTION:
This is a Phase 2, multicentre, multinational, randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of two intravenous (IV) treatment regimens of anifrolumab versus placebo while taking standard of care (SOC) treatment with mycophenolate mofetil (MMF) and corticosteroids in adult subjects with active proliferative lupus nephritis (LN).

ELIGIBILITY:
Main Inclusion Criteria:

1. Age 18 through 70 years at the time of screening
2. Fulfils at least 4 of the 11 criteria of the revised 1982 ACR classification criteria for SLE, at least one of which must be:

   1. Positive antinuclear antibody (ANA) test (1:40 or higher) or
   2. Elevated anti-dsDNA antibodies at screening (reported as equivocal or positive results), as per the centrallaboratory; or
   3. Anti-Smith antibody at screening elevated to above normal (ie, positive or equivocal results) as per the central laboratory
3. Class III (±Class V) or Class IV (±Class V) LN according to the World Health Organisation (WHO) or 2003 ISN/RPS classification based on a renal biopsy obtained within 12 weeks prior to signing the ICF or during the screening period:
4. Urine protein to creatinine ratio >1 gm/gm (113.17 mg/mmol), obtained on a 24-hour urine collection at screening
5. Estimated glomerular filtration rate ≥35 mL/min/1.73 m2
6. Must not have active or latent TB on either chest radiograph or by Quantiferon gold test
7. Women of childbearing potential must have a negative serum beta-hCG test at screening and negative urine pregnancy test prior to the first dose of sponsor-provided MMF.

Main Exclusion Criteria:

1. Receipt of any investigational product (small molecule or biologic) or commercially available biologic agent within four weeks or 5 half lives prior to signing of the ICF, whichever is greater
2. Pure Class V membranous LN on a renal biopsy obtained within 12 weeks prior to signing ICF or during the screening period
3. Known intolerance to ≤1.0 gm/day of MMF
4. History of dialysis within 12 months prior to signing the ICF or expected need for renal replacement therapy (dialysis or renal transplant) within a 6 month period after enrolment
5. Subjects, who at the time of signing the ICF, received any of the following immunosuppressive therapies after their qualifying biopsy

   1. Oral corticosteroids >0.5 mg/kg/day for more than 8 weeks or
   2. Oral or IV pulse methylprednisolone >3.0 gm (cumulative dose) or
   3. IV cyclophosphamide >2 pulses of high-dose (≥0.5 gm/m2) or >4 doses of low dose (500 mg every 2 weeks) or
   4. Average MMF >2.5 gm/day (>1800 mg/day of enteric-coated mycophenolate sodium) for more than 8 weeks or
   5. Tacrolimus >4 mg/day for more than 8 weeks
6. Major surgery within 8 weeks before signing the ICF or major surgery planned during the study period
7. History of any non-SLE disease that has required treatment with oral or parenteral corticosteroids for more than a total of 2 weeks within the last 24 weeks prior to signing the ICF
8. Confirmed positive test for hepatitis B or hepatitis C
9. Any severe herpes infection at any time prior to randomization
10. Opportunistic infection requiring hospitalisation or parenteral antimicrobial treatment within 3 years prior to randomization (vaginal, oral and skin candidiasis is not an exclusionreason).
11. History of cancer, apart from:

    1. Squamous or basal cell carcinoma of the skin that has been successfully treated
    2. Cervical cancer in situ that has been successfully treated
12. Concurrent enrolment in another clinical study with an IP within 4 weeks prior to ICF signing or within 5 half-lives of the IP used in that clinical study, whichever is longer.
13. During screening (within 30 days before Day 1 [Week 0 visit]), any of the following:

    1. Aspartate transaminase (AST) >2.5×upper limit of normal (ULN)
    2. Alanine transaminase (ALT) >2.5×ULN
    3. Total bilirubin >ULN (unless due to Gilbert's syndrome [based on Investigator's judgement])
    4. Glycosylated haemoglobin (HbA1c) >8% (or >0.08) at screening (diabetic subjects only)
    5. Neutrophil count <1x103/μL (or <1.0 GI/L)
    6. Platelet count <25x103/μL (or <25 GI/L)
    7. Haemoglobin <8 g/dL (or <80 g/L).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AB, Study Director — AstraZeneca
Locations (65):
- United States (16):
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Thousand Oaks, California
  - Research Site, Aurora, Colorado
  - Research Site, DeBary, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Newark, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Memphis, Tennessee
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Rosario
- Australia (4):
  - Research Site, Adelaide
  - Research Site, Clayton
  - Research Site, Parkville
  - Research Site, Westmead
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- France (5):
  - Research Site, Bordeaux
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (2):
  - Research Site, Berlin
  - Research Site, Kiel
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
  - Research Site, Szeged
- Italy (4):
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Reggio Emilia
- Mexico (4):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, San Luis Potosí City
- Peru (2):
  - Research Site, Arequipa
  - Research Site, Lima
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Orenburg
  - Research Site, Saint Petersburg
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Niš
  - Research Site, Novi Sad
- South Korea (3):
  - Research Site, Gwangju
  - Research Site, Seoul
  - Research Site, Suwon
- Research Site, Barcelona, Spain
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Jayne D, Rovin B, Mysler E, Furie R, Houssiau F, Trasieva T, Knagenhjelm J, Schwetje E, Tang W, Tummala R, Lindholm C. Anifrolumab in lupus nephritis: results from second-year extension of a randomised phase II trial. Lupus Sci Med. 2023 Aug;10(2):e000910. doi: 10.1136/lupus-2023-000910. PMID 37607780
- [Derived] Jayne D, Rovin B, Mysler EF, Furie RA, Houssiau FA, Trasieva T, Knagenhjelm J, Schwetje E, Chia YL, Tummala R, Lindholm C. Phase II randomised trial of type I interferon inhibitor anifrolumab in patients with active lupus nephritis. Ann Rheum Dis. 2022 Apr;81(4):496-506. doi: 10.1136/annrheumdis-2021-221478. Epub 2022 Feb 10. PMID 35144924
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00007&attachmentIdentifier=91395ece-af3d-4a03-b57b-c464aaf45d6a&fileName=PXL_221659_D3461C00007_protocol_Redacted_FINAL.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00007&attachmentIdentifier=8fbb335e-c784-4c5f-b9e6-72b7d71c2c34&fileName=PXL_221659_D3461C00007_SAP_redacted_Redacted_FINAL.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00007&attachmentIdentifier=52b710e6-cca2-41c8-ac3f-457b0c728df5&fileName=PXL_221659_D3461C00007_Clinical_Study_Report_Synopsis_Final_Redacted_FINAL.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were randomized at 66 sites in 16 countries. The study was conducted from 04 November 2015 to 18 January 2021.
Pre-assignment Details: The screening period was from Day -30 to Day -1. Informed consent form (ICF) was signed prior to screening procedures. All the study assessments were performed as per the schedule of assessment.
Groups:
- Anifrolumab - Basic Regimen: Subjects were administered with lower dose of Anifrolumab intravenously (IV) every 4 weeks (Q4W) from Week 0 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
- Anifrolumab - Intensified Regimen: Subjects were administered with higher dose of Anifrolumab IV Q4W for first 3 doses followed by lower dose from Week 12 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
- Placebo: Subjects were administered with placebo every 4 week from Week 0 to Week 100 in addition to SOC which continued until Week 112.
Period: Overall Study
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | Placebo
Started | 46 | 52 | 49
FAS (Full Analysis Set) (Patients did not receive IP) | 45 | 51 | 49
Completed | 18 | 28 | 20
Not Completed | 28 | 24 | 29
Not completed — Withdrawal by Subject | 9 | 6 | 10
Not completed — Adverse Event | 3 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 5 | 7 | 4
Not completed — Death | 1 | 0 | 0
Not completed — Non-responding completer, Not eligible for extension study, Use of any restricted Medications | 4 | 8 | 9
Not completed — TECHNICAL PROBLEMS | 1 | 0 | 0
Not completed — PROGRESSIVE DISEASE | 1 | 0 | 2
Not completed — Physician Decision | 2 | 1 | 2
Not completed — Patients did not receive IP | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all subjects who received at least one dose of study treatment and were analyzed according to randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | Placebo | Total
Number analyzed (Participants) | 45 | 51 | 49 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (11.49) | 35.0 (10.58) | 34.0 (10.18) | 34.7 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 45 | 38 | 120
  Male | 8 | 6 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 20 | 65
  Not Hispanic or Latino | 23 | 28 | 29 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 0 | 4
  Asian | 11 | 7 | 10 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 4 | 1 | 7
  White | 17 | 25 | 24 | 66
  Other | 11 | 14 | 14 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Urine Protein to Creatinine Ratio (UPCR)
Description: To evaluate the efficacy of anifrolumab plus SOC (combination of mycophenolate mofetil and corticosteroids) compared with placebo plus SOC in subjects with active proliferative lupus nephritis (LN).
  Geometric mean ratio of 24-hour UPCR at week 52 over baseline. Values <1 indicate improvement from baseline.
Time Frame: From Week 1 (Baseline) up to Week 52
Population: Full analysis set (FAS): The FAS included all subjects who received at least one dose of study treatment and were analyzed according to randomized treatment (mITT principle).
  Here, overall number of subjects analyzed signifies the subjects with available data that were analyzed for the outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: milligram/milligram (mg/mg)
Groups:
- All Anifrolumab: This arm comprises Anifrolumab - Basic Regimen and Anifrolumab - Intensified Regimen.
  Anifrolumab - Basic Regimen: Subjects were administered with lower dose of Anifrolumab intravenously (IV) every 4 weeks (Q4W) from Week 0 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
  Anifrolumab - Intensified Regimen: Subjects were administered with higher dose of Anifrolumab IV Q4W for first 3 doses followed by lower dose from Week 12 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | All Anifrolumab | Placebo
Number analyzed (Participants) | 41 | 50 | 91 | 41
milligram/milligram (mg/mg) | 0.326 [0.190 to 0.561] | 0.285 [0.177 to 0.457] | 0.305 [0.198 to 0.468] | 0.296 [0.175 to 0.499]
Statistical Analysis 1: Comparison: All Anifrolumab vs Placebo; The model includes fixed effects for treatment group, visit, stratification factors, log-transformed 24-hour UPCR at baseline, and treatment-by-visit interaction. All data up to and including the date of discontinuation of study treatment were included in the analysis; Test type: Superiority; p = 0.9052, Mixed Models Analysis — The p-values presented are unadjusted and was compared with the respective adjusted significance level (α). If α is not displayed, no formal testing can be performed and the corresponding p-value was nominal; Geometric Mean Ratio = 1.031, 95% CI 2-sided [0.621 to 1.713] — Geometric mean ratio >1 favours placebo

2. Secondary Outcome: Proportion of Subjects Achieving the Composite Endpoint Complete Renal Response (CRR)
Description: CRR was defined as meeting all of the following:
  * Estimated glomerular filtration rate (eGFR) is ≥60 mL/min/1.73 m^2 or no confirmed decrease of eGFR from baseline of ≥20%
  * 24-hour UPCR ≤ 0.7 mg/mg
  * No discontinuation of investigational product (IP) or use of restricted medication beyond the protocol allowed threshold before assessment
  * eGFR was based on Modification of Diet in Renal Disease (MDRD) formula. Subjects treated with restricted medication beyond the protocol allowed threshold, or discontinuing study treatment for other reasons, were regarded as non-responders.
Time Frame: Week 52
Population: The FAS included all subjects who received at least one dose of study treatment and were analyzed according to randomized treatment (mITT principle). The subjects being analyzed was less than the number of patients in the FAS. Subjects from France and Italy were excluded from the analysis (France EC and Italy HA did not accept CSP amendment 3 (version 4.0)).
Measure: Number; unit: Percentage of subjects
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | All Anifrolumab | Placebo
Number analyzed (Participants) | 45 | 51 | 96 | 49
Percentage of subjects
  Responder: number analyzed (Participants) | 43 | 44 | 87 | 45
  Responder | 16.3 | 45.5 | 31.0 | 31.1
  Non-responder: number analyzed (Participants) | 43 | 44 | 87 | 45
  Non-responder | 83.7 | 54.5 | 69.0 | 68.9
Statistical Analysis 1: Comparison: All Anifrolumab vs Placebo; The statistical analysis represents the estimated percentage of responders. The responder/non-responder rates (percentages), the difference in estimates and associated 95% CI are weighted and are calculated using a stratified Cochran-Mantel-Haenszel (CMH) approach; Test type: Superiority; p = 0.9929, Cochran-Mantel-Haenszel — At Week 52, the p-values presented are unadjusted and will be compared to the respective adjusted significance level (α). If α is not displayed no formal testing can be performed and the corresponding p-value is nominal; Difference in estimates = -0.08, 95% CI 2-sided [-16.92 to 16.76]

3. Other Pre Specified Outcome: Number of Subjects With Adverse Events
Description: To assess AEs (non-serious, serious and adverse event of special interest (AESI)) as variables of safety and tolerability of anifrolimab.
  The AESIs are serious infections, including non-opportunistic serious infections, opportunistic infections, anaphylaxis, malignancy, herpes zoster, TB (including latent TB), influenza, vasculitis (non-SLE), and MACE (including stroke, acute coronary syndrome, myocardial infarction, or cardiovascular death).
  Study period: During treatment and follow-up data are presented.
Time Frame: From screening (Day-30 to -1) period until the follow-up period (Week 112)
Population: Full analysis set (FAS): The FAS included all subjects who received at least one dose of study treatment and were analyzed according to randomized treatment (mITT principle).
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | All Anifrolumab | Placebo
Number analyzed (Participants) | 45 | 51 | 96 | 49
Participants
  Subjects with any AE- During treatment | 43 | 47 | 90 | 44
  Subjects with any acute AE- During treatment | 11 | 15 | 26 | 14
  Any AE with outcome of death- During treatment | 0 | 0 | 0 | 0
  Any SAE (including events with- outcome of death)- During treatment | 10 | 9 | 19 | 8
  Any AE leading to discontinuation of investigational product- During treatment | 5 | 6 | 11 | 5
  Any AE related to investigational product (investigator assessment)- During treatment | 24 | 13 | 37 | 16
  Any AE of severe intensity- During treatment | 6 | 7 | 13 | 8
  Any AESI- During treatment | 12 | 12 | 24 | 8
  Non-opportunistic serious infections- During treatment | 0 | 1 | 1 | 3
  Opportunistic infections- During treatment | 1 | 0 | 1 | 1
  Anaphylaxis- During treatment | 0 | 0 | 0 | 0
  Malignancy- During treatment | 0 | 1 | 1 | 0
  Herpes zoster- During treatment | 9 | 7 | 16 | 4
  Tuberculosis/LTB (latent tuberculosis)- During treatment | 0 | 0 | 0 | 0
  Influenza- During treatment | 2 | 4 | 6 | 1
  Vasculitis (non-systemic lupus erythematosus)- During treatment | 0 | 0 | 0 | 0
  Major adverse cardiovascular events according to the CV-EAC- During treatment | 0 | 0 | 0 | 1
  Any other significant AE- During treatment | 0 | 0 | 0 | 0
  Subjects with any AE- follow-up | 12 | 8 | 20 | 22
  Any AE with outcome of death- follow-up | 1 | 0 | 1 | 0
  Any SAE (including events with outcome of death)- follow-up | 3 | 0 | 3 | 3
  Any AE related to investigational product (investigator assessment)- follow-up | 2 | 0 | 2 | 1
  Any AE of severe intensity- follow-up | 2 | 0 | 2 | 3
  Any AESI- follow-up | 2 | 0 | 2 | 2
  Non-opportunistic serious infections- follow-up | 0 | 0 | 0 | 1
  Opportunistic infections- follow-up | 0 | 0 | 0 | 0
  Anaphylaxis- follow-up | 0 | 0 | 0 | 0
  Malignancy- follow-up | 0 | 0 | 0 | 0
  Herpes zoster- follow-up | 2 | 0 | 2 | 1
  Tuberculosis/LTB- follow-up | 0 | 0 | 0 | 0
  Influenza- follow-up | 0 | 0 | 0 | 0
  Vasculitis (non-SLE)- follow-up | 0 | 0 | 0 | 0
  Major adverse cardiovascular events according to the CV-EAC- follow-up | 0 | 0 | 0 | 0
  Any other significant AE- follow-up | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Number of Subjects With Suicidal Ideation and Behavior and Suicide Attempts Via Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS was used to assess the suicidal ideation and behavior and suicide attempts on a graded scale from 1 to 5. 1 indicates as low suicidal and 5 as high suicidal behavior.
Time Frame: Baseline, treatment and follow up (an average of 60 weeks)
Population: Full analysis set (FAS): The FAS included all subjects who received at least one dose of study treatment and were analyzed according to randomized treatment (mITT principle).
  Here, number analyzed in each row signifies only the subjects with available data that were analyzed for each parameter/ timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | All Anifrolumab | Placebo
Number analyzed (Participants) | 45 | 51 | 96 | 49
Participants
  Suicidal attempts: Baseline: number analyzed (Participants) | 44 | 50 | 94 | 48
  Suicidal attempts: Baseline | 0 | 0 | 0 | 0
  Suicidal attempts: Treatment: number analyzed (Participants) | 45 | 51 | 96 | 47
  Suicidal attempts: Treatment | 0 | 0 | 0 | 0
  Suicidal attempts: Follow up: number analyzed (Participants) | 17 | 18 | 35 | 23
  Suicidal attempts: Follow up | 0 | 0 | 0 | 0
  Suicidal behaviour: Baseline | 0 | 0 | 0 | 0
  Suicidal behaviour: Treatment | 0 | 0 | 0 | 0
  Suicidal behaviour: Follow up | 0 | 0 | 0 | 0
  Suicidal ideation: Baseline | 0 | 2 | 2 | 4
  Suicidal ideation: Treatment | 0 | 0 | 0 | 2
  Suicidal ideation: Follow up | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: Total Score of Personal Health Questionnaire Depression Scale-8 (PHQD-8)
Description: PHQ-8 is a 8-item self-report scale, all items are rated on a score of 0-3, for a total range of 0-24. PHQ-8 assesses symptoms of depression over the previous 2 weeks. Higher scores indicate more depressive symptoms.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 52, Week 60
Population: Full analysis set (FAS): The FAS included all subjects who received at least one dose of study treatment and were analyzed according to randomized treatment (mITT principle).
  Here, number analyzed in each row signifies only the subjects with available data that were analyzed for each timeframe.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | All Anifrolumab | Placebo
Number analyzed (Participants) | 45 | 51 | 96 | 49
Score on a scale
  Baseline: number analyzed (Participants) | 43 | 51 | 94 | 46
  Baseline | 5.1 (4.34) | 4.3 (4.05) | 4.6 (4.18) | 5.8 (4.54)
  Week 12: number analyzed (Participants) | 36 | 50 | 86 | 41
  Week 12 | 3.4 (3.88) | 3.1 (3.56) | 3.2 (3.68) | 5.1 (4.84)
  Week 24: number analyzed (Participants) | 36 | 48 | 84 | 42
  Week 24 | 2.7 (2.41) | 2.5 (3.18) | 2.6 (2.86) | 4.9 (5.10)
  Week 36: number analyzed (Participants) | 38 | 42 | 80 | 40
  Week 36 | 3.3 (4.04) | 2.5 (3.22) | 2.8 (3.63) | 3.5 (2.73)
  Week 52: number analyzed (Participants) | 29 | 35 | 64 | 35
  Week 52 | 2.3 (3.44) | 3.4 (5.24) | 2.9 (4.51) | 4.2 (3.30)
  Week 60: number analyzed (Participants) | 6 | 8 | 14 | 5
  Week 60 | 3.3 (4.80) | 5.6 (7.01) | 4.6 (6.06) | 4.6 (2.07)

6. Other Pre Specified Outcome: Extra-renal Flares Using Systemic Lupus Erythematosus (SLE) Disease Activity Index 2000 (SLEDAI 2K) Based Flare Assessment Instrument
Description: Flare will be defined as any one criterion present in either the Mild/Moderate Flare and/or Severe Flare categories. New or worsened manifestation should only be reported for manifestations of SLE. The SLEDAI-2K score range is 0 to 105 with higher scores representing increased disease activity.
  Mild/ Moderate flare defined as change in non-renal components of the SLEDAI-2K instrument score of ≥3 but <7 points compared to previous visit. Severe Flare defined as change in non-renal components of the SLEDAI-2K instrument score by ≥7 points compared to previous visit.
  The flare rate per subject year is defined as the number of subjects with a respective flare divided by the sum of exposure time in days for all subjects in the analysis set multiplied by 365.25.
Time Frame: From baseline up to week 112
Population: Full analysis set (FAS): The FAS included all subjects who received at least one dose of study treatment and were analyzed according to randomized treatment (mITT principle).
  Here, number analyzed in each row signifies only the subjects with available data that were analyzed for each parameter
Measure: Number; unit: Flare rate per subject year
Arm/Group | Anifrolumab - Basic Regimen | Anifrolumab - Intensified Regimen | All Anifrolumab | Placebo
Number analyzed (Participants) | 45 | 51 | 96 | 49
Flare rate per subject year
  Mild/moderate: All flares | 0.019 | 0.016 | 0.017 | 0.016
  Mild/moderate: On-treatment | 0.017 | 0.012 | 0.014 | 0.010
  Mild/moderate: Off-treatment | 0.002 | 0.003 | 0.003 | 0.006
  Severe: All flares | 0.007 | 0.001 | 0.003 | 0.006
  Severe: On-treatment | 0.004 | 0.00 | 0.002 | 0.004
  Severe: Off-treatment | 0.003 | 0.001 | 0.002 | 0.002

ADVERSE EVENTS:
Time Frame: From screening (Day-30 to -1) period until follow-up (Week 112).
Groups:
- Anifrolumab - Basic Regimen- Treatment Period; Anifrolumab - Basic Regimen- Follow up: Subjects were administered with lower dose of Anifrolumab intravenously (IV) every 4 weeks (Q4W) from Week 0 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
- Anifrolumab - Intensified Regimen- Treatment Period; Anifrolumab - Intensified Regimen- Follow up: Subjects were administered with higher dose of Anifrolumab IV Q4W for first 3 doses followed by lower dose from Week 12 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
- All Anifrolumab- Treatment Period; All Anifrolumab- Follow up: This arm comprises Anifrolumab - Basic Regimen and Anifrolumab - Intensified Regimen.
  Anifrolumab - Basic Regimen: Subjects were administered with lower dose of Anifrolumab intravenously (IV) every 4 weeks (Q4W) from Week 0 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
  Anifrolumab - Intensified Regimen: Subjects were administered with higher dose of Anifrolumab IV Q4W for first 3 doses followed by lower dose from Week 12 to Week 100, in addition to pre-specified standard of care (SOC) which continued until Week 112.
- Placebo- Treatment Period; Placebo- Follow up: Subjects were administered with placebo every 4 week from Week 0 to Week 100 in addition to SOC which continued until Week 112.
Arm/Group | Anifrolumab - Basic Regimen- Treatment Period | Anifrolumab - Intensified Regimen- Treatment Period | All Anifrolumab- Treatment Period | Placebo- Treatment Period | Anifrolumab - Basic Regimen- Follow up | Anifrolumab - Intensified Regimen- Follow up | All Anifrolumab- Follow up | Placebo- Follow up
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/51 | 0/96 | 0/49 | 1/45 | 0/51 | 1/96 | 0/49
Serious Adverse Events (participants affected / at risk) | 10/45 | 9/51 | 19/96 | 8/49 | 3/45 | 0/51 | 3/96 | 3/49
Other Adverse Events (participants affected / at risk) | 31/45 | 39/51 | 70/96 | 33/49 | 0/45 | 0/51 | 0/96 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anifrolumab - Basic Regimen- Treatment Period (N=45) | Anifrolumab - Intensified Regimen- Treatment Period (N=51) | All Anifrolumab- Treatment Period (N=96) | Placebo- Treatment Period (N=49) | Anifrolumab - Basic Regimen- Follow up (N=45) | Anifrolumab - Intensified Regimen- Follow up (N=51) | All Anifrolumab- Follow up (N=96) | Placebo- Follow up (N=49)
Herpes zoster (Infections and infestations) | 3 | 3 | 6 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Abscess bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Varicella zoster pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Histoplasmosis disseminated (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lupus endocarditis (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anifrolumab - Basic Regimen- Treatment Period (N=45) | Anifrolumab - Intensified Regimen- Treatment Period (N=51) | All Anifrolumab- Treatment Period (N=96) | Placebo- Treatment Period (N=49) | Anifrolumab - Basic Regimen- Follow up (N=45) | Anifrolumab - Intensified Regimen- Follow up (N=51) | All Anifrolumab- Follow up (N=96) | Placebo- Follow up (N=49)
Urinary tract infection (Infections and infestations) | 10 | 6 | 16 | 5 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 9 | 15 | 9 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 7 | 15 | 8 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 7 | 11 | 6 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 6 | 4 | 10 | 4 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 4 | 7 | 2 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 3 | 6 | 2 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 3 | 2 | 5 | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 4 | 5 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 5 | 4 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7 | 4 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 7 | 10 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 5 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 4 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 4 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The submission/document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT02547922/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT02547922/SAP_001.pdf